CLINICAL TRIAL: NCT06319378
Title: CAPSI - Cancer Related Major Depression Treated With a Single Dose of Psilocybin: A Multicenter Randomized Placebo Controlled Double Blind Clinical Trial
Brief Title: Cancer Related Major Depression Treated With a Single Dose of Psilocybin
Acronym: CAPSI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Section for Affective Disorders; Northern Stockholm Psychiatry (Other)
Collaborators: Uppsala University Hospital (Other); Region Örebro County (Other); Vastra Gotaland Region (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPSI no 2 date 231024; 2023-505532-35-00 (Other: CTIS)
Record Dates: First submitted 2023-11-08; First posted 2024-03-20 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: MDD
Keywords: malignant neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Psilocybin; Superoxide Dismutase

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, active placebo, randomization ratio 2:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psilocybin 25 mg (active) (Experimental)
  Interventions: Drug: psilocybin 25 mg sod
- psilocybin 1 mg (Active Comparator)
  Interventions: Drug: psilocybin 1 mg sod

INTERVENTIONS:
Drug: psilocybin 25 mg sod — psilocybin 25 mg sod
  Arms: psilocybin 25 mg (active)
Drug: psilocybin 1 mg sod — active placebo
  Arms: psilocybin 1 mg

SUMMARY:
The goal of this randomized placebo controlled trial is to compare the antidepressant effect of a single oral dose of psilocybin 25 mg compared to 1 mg in 100 patients with cancer related major depressive disorder. The main question it aims to answer is:

The primary objective of this study is to evaluate the efficacy of a single 25 mg oral dose of psilocybin for major depressive disorder (MDD) compared to an active placebo (psilocybin 1 mg) assessed as the difference between groups in changes in depressive symptoms, in the following Population: 20-80 (inclusive) years old, current depressive episode (according to Patient Health Questionnaire (PHQ-9)

≥10), >1 month after cancer diagnosis, with at least 12 months of life expectancy, willingness to abstain from other psychotherapeutic or antidepressant treatments during the study (wash out time 5 half-lives).

ELIGIBILITY:
Inclusion Criteria

* signed informed consent via minavårdkontakter.se
* Are 20 to 80 (inclusive) years old at the time of signed informed consent
* Are able to read, speak, and understand Swedish
* Are able and willing to adhere to study requirements, including attending all study visits, preparatory and follow-up sessions, and completing all study evaluations
* Are able to swallow capsules
* Women of childbearing potential (WOCBP) must agree to practice an effective means of birth control throughout the duration of exposure to the Investigational Product, from Screening through the Day 8.
* A diagnosis of a malignant neoplasm with a diagnostic code from C00 to C97 according to the International Classification of Diseases and Related Health Problems, 10th Revision (ICD-10)
* ≥1 month after cancer diagnosis and ≥ 12 months of life expectancy at time of inclusion
* physical functioning performance status 0-2 (World Health Organisation/Eastern Cooperative Oncology Group (WHO/ECOG))
* Meet ICD-10 criteria for a diagnosis of major depressive disorder and are currently experiencing a major depressive episode of at least a 30-day duration at the time of the Screening less than 1 year at time of Screening
* Have moderate-severe depression symptoms at Screening, as defined by a Screening PHQ-9 total score ≥ 10.
* Are willing to abstain from other psychotherapeutic or antidepressant treatments during the study period (180 days; wash out time 5 half-lives). Note, if antidepressant treatment becomes needed as determined by the study physician this will be supported by the study personnel.
* Have an identified support person.
* Agree to be driven/accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing

Exclusion Criteria

* Individuals not eligible to be randomized in this protocol are those who meet any of the following criteria:
* Last contact with health care due to cancer monitoring or treatment >1 year ago.
* Women who are pregnant, as indicated by a positive urine pregnancy test at Screening or Baseline. Women who intend to become pregnant during the study or who are currently nursing.
* Unwilling or unable to discontinue formal psychotherapy
* Ongoing antidepressant drug treatment. No interruption of ongoing antidepressant treatment will be done on the initiation of the study personnel. Patients will be encouraged to discuss any interruption with their responsible clinical physician.
* Have previously during the current episode received the following non-medication treatments: deep brain stimulation (DBS); vagus nerve stimulation (VNS)
* Currently receiving electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS)
* Unable or unwilling to discontinue any current medications that are known uridine diphosphate (UDP) or glucuronosyltransferase (UGT) enzyme modulators (eg valproate) Note: Any prohibited agents must have been stopped at least 5x the elimination half-life of the specific drug plus one week at the time of Baseline. See Appendix A for a full list of prohibited medications.
* Report psychedelic substances use ever

  o Note: Psychedelic substances include psilocybin, Lysergic acid diethylamide (LSD), mescaline (and natural products containing mescaline including peyote and San Pedro cactus), N,N-Dimethyltryptamine (DMT), natural products containing DMT including ayahuasca and 5-Methoxy-N,N-dimethyltryptamine (5-MeO-DMT), ibogaine, 3,4-methylenedioxy- methamphetamine (MDMA) or other psychedelics.
* Cancer at time of inclusion involving the Central Nervous System (CNS) (as determined by a clinical examination or Magnetic Resonance Imaging (MRI))
* Cancer treatment/follow up regime determined to be incompatible with the CAPSI protocol (eg due to time lines, interaction between cancer treatment and psilocybin 25 mg or 1 mg exposure).
* Have any of the following cardiovascular conditions:

  * congenital long QT syndrome (prior diagnosis),
  * any of the following if disabling physical exercise similar to walking two stairs without pause: coronary artery disease, cardiac hypertrophy, cardiac ischemia, congestive heart failure
  * a clinically significant Screening Electro Cardio-Graphy (ECG) abnormality (e.g., atrial fibrillation);
  * artificial heart valve; or
  * any other significant current or history of cardiovascular condition, based on the clinical judgment of study physician, that would make a participant unsuitable for the study
* At Screening or Baseline have elevated blood pressure as defined as:

  a. Screening blood pressure Systolic Blood Pressure >150 mmHg or Diastolic Blood Pressure > 95 mmHg on three separate readings; or

  o Baseline blood pressure SBP >160 mmHg or DBP > 100 mmHg on three separate readings
* Have a history of stroke or Transient Ischemic Attack (TIA)
* Have moderate to severe hepatic impairment, as indexed by a Child-Pugh score ≥ 7
* Have uncontrolled epilepsy
* Have insulin-dependent diabetes
* Note: Participants who are taking oral hypoglycemic agent and have a history of hypoglycemia requiring medical intervention will be excluded
* Are unable or unwilling to adhere to the following medication requirements:
* Agree to suspend sildenafil (Viagra®), tadalafil, or similar medications at least 72 hours prior to dosing
* Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Cannabis, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP), and Tetrahydrocannabinol (THC). Exceptions are made for prescribed Benzodiazepines (stable dose for sleep or anxiety).

  o Note: Benzodiazepine medications for sleep and non-benzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for at least 6 weeks prior to Screening, as determined during review of concomitant medications Note: Participants using cannabis, including legal cannabis, for any purposes will be excluded Note: Participants who are taking prescription maintenance methadone or buprenorphine naloxone will be excluded Note: Prescription opiates must have been stopped at least 5x the elimination half- life of the specific drug at the time of inclusion, as confirmed with a negative urine drug screen.
* Nicotine dependence that would disallow an individual to be nicotine free for the 7-10 hours during the dosing period
* Meet International Classification of Diseases version 10 (ICD-10) criteria for schizophrenia spectrum or other psychotic disorders, including MDD with psychotic features (except substance/medication-induced or due to another medical condition), or Bipolar I Disorder, Bipolar II Disorder.

Note: Participants with any lifetime diagnosis of schizophrenia spectrum or other psychotic disorders will be excluded

* Meet ICD-10 criteria for antisocial personality disorder
* Meet ICD-10 criteria for a moderate or severe alcohol or drug use disorder (excluding caffeine) Note: Participants with a diagnosis of alcohol or drug use disorder within the past 12 months will be excluded
* Have the presence of any psychiatric condition or symptom judged by the PI (or designee) to be a more significant clinical problem than MDD for the participant.
* Have a first-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition).
* Have a psychiatric condition judged to be incompatible with establishment of rapport with the Facilitators or safe exposure to psilocybin
* Report the following suicidal ideation or suicidal thoughts defined as

  * Have a score of ≥ 5 on Item 10 (suicidal thoughts) on MADRS at Screening or Baseline; or
  * Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior at any time prior to randomization
  * Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior
* Have any physical or psychological symptom, medication or other relevant finding at Screening or Baseline, based on the clinical judgment of clinical/medical study personnel, that would make a participant unsuitable for the study.
* Have an allergy or intolerance to any of the materials contained in either drug product
* Have Hepatitis B, C or HIV (HIV only allowed if on treatment and non-detectable virus
* concentrations)
* Have one or more clinically relevant pathological blood test results (as determined by a study physician; with the exception of CRP).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-17 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MADRS at day 42 | day 42
  Montgomery Asberg Depression Rating Scale (MADRS) total score (0-60, smaller equals better)

SECONDARY OUTCOMES:
MADRS day 8 | day 8
  Montgomery Asberg Depression Rating Scale (MADRS) total score (0-60, smaller equals better)
MADRS-S at all evaluations between Day 0 and Day 42 (Mixed Models for Repeated Measures (MMRM) x1) | Day 42
  Montgomery Asberg Depression Rating Scale self rating (MADRS-S) (0-54, smaller equals better)
SDS at Day 42 | Day 42
  Sheehan Disability Scale (SDS) (0-10, smaller equals better)
CGI at Day 8 and Day 42 (analysis of covariance (ANCOVA) x6) | Day 8 and 42
  Clinical Global Impression (CGI), (1-7, smaller equals better)
EQ-5D-5L at Day 8 and Day 42 (ANCOVA x6) | Day 8 and 42
  Euroquol 5 Dimension scale (EQ5D-5L), 0-1, higher equals better
AQOL-6D at Day 42 (ANCOVA x1) | Day 42
  Assessing Quality of Life 6 dimensions (AQOL-6D) (0-99, smaller equals better)
MADRS at Day 90 and Day 180 (ANCOVA x2) | Day 90 and Day 180
  Montgomery Asberg Depression Rating Scale (MADRS) total score (0-60, smaller equals better)
MADRS-S at all evaluations between Day 43 and Day 180 (MMRM x1) | between Day 43 and Day 180
  Montgomery Asberg Depression Rating Scale self rating (MADRS-S) (0-54, smaller equals better)
SDS at Day 180 (ANCOVA x3) | Day 180
  Sheehan Disability Scale (SDS) (0-10, smaller equals better)
GAD-7 at Day 180 (ANCOVA x3) | Day 180
  General Anxiety Disorder 7 (GAD-7) (0-21, lower equals better)
HADS at Day 180 (ANCOVA x3) | Day 180
  Hospital Anxiety and Depression Scale (HADS) (0-42, smaller equals better)
CGI at Day 90 and Day 180 (ANCOVA x6) | Day 90 and Day 180
  Clinical Global Impression (CGI), (1-7, smaller equals better)
EQ-5D-5L at Day 90 and Day 180 (ANCOVA x6) | Day 90 and Day 180
  Euroqol 5 Dimension scale (EQ5D-5L), 0-1, higher equals better
AQOL-6D at Day 90 and Day 180 (ANCOVA x2) | Day 90 and Day 180
  Assessing Quality of Life 6 dimensions (AQOL-6D) (0-99, smaller equals better)
GAD-7 at Day 42 | Day 42
  General Anxiety Disorder 7 (GAD-7) (0-21, lower equals better)
HADS at Day 42 | Day 42
  Hospital Anxiety and Depression Scale (HADS) (0-42, smaller equals better)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Lundberg, MD PhD, Principal Investigator — Norra Stockholms Psykiatri and Karolinska Institutet
Locations (4):
- Sweden (4):
  - region Västra Götaland, Gothenburg
  - Örebro sjukhus, Örebro
  - Norra Stockholms Psykiatri, Stockholm
  - Psykiatriska Kliniken, Akademiska Sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://ki.se/en/cns/capsi